CLINICAL TRIAL: NCT07131215
Title: Smart Technology-Based Intervention and Monitoring of Physical and Mental Health in Early Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YI-JU TSAI (Other)
Responsible Party: Sponsor-Investigator, YI-JU TSAI, Professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCKU_Postmenopausal
Record Dates: First submitted 2025-07-20; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Postmenopausal; Postmenopausal Disorder; Menopause
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- APP exercise group (Experimental): 8-week home-based multimodal exercise program via customized mobile APP
  Interventions: Other: Home-based multimodal exercise; Other: Education
- Supervised exercise group (Experimental): 8-week supervised exercise program in the laboratory
  Interventions: Other: Supervised multimodal exercise program; Other: Education
- Education control group (Other): 30-minute educational session
  Interventions: Other: Education

INTERVENTIONS:
Other: Home-based multimodal exercise — Mobile Applications
  Arms: APP exercise group
Other: Supervised multimodal exercise program — In laboratory
  Arms: Supervised exercise group
Other: Education — Menopause education

SUMMARY:
The aim of this study is to compare the short-term and long-term effects of an 8-week home-based multimodal exercise program, delivered through a smartphone app, on quality of life, muscle function, and physical performance in early postmenopausal women.

DETAILED DESCRIPTION:
The goal of this study is to investigate whether a comprehensive exercise program in early postmenopause can improve quality of life, physical function, and long-term health.

The main question it aims to answer is:

Does adding exercise intervention in early postmenopause will improve their quality of life and long-term health?

ELIGIBILITY:
Inclusion Criteria:

* 45 to 65-year-old postmenopausal women
* At least 12 months of amenorrhea
* Within 6 years after menopause

Exclusion Criteria:

* Exercised more than twice a week for at least 30 minutes per session
* Received hormone therapy in the past three months
* Neurological disease (e.g., spinal cord injury, multiple sclerosis, stroke) or cardiovascular diseases
* History of pelvic or prolapse surgery (excluding cesarean section)
* History of malignancy affecting the bladder, urethra, uterus, ovary, cervix, or rectum
* Using medications that could affect heart rate or mood
* Body mass index (BMI) > 35 kg/m²

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle function measures for lumbopelvic muscle: Abdominal and back muscles | Changes from baseline to 8 weeks when participants finish the intervention.
  Ultrasonography images of muscle thickness of abdominal and back muscles during rest and during active straight leg raise. Each condition will be tested three times. Muscle thickness at rest and during contraction will be measured using ImageJ, with results expressed in millimeters (mm)
Muscle function measures for lumbopelvic muscle | Changes from baseline to 8 weeks when participants finish the intervention.
  Ultrasonography images of bladder displacement for pelvic floor muscles during rest, maximum contraction, and during active straight leg raise. Each condition will be tested three times. Bladder height differences between contraction and relaxation of the pelvic floor muscles will be measured using ImageJ, with results expressed in millimeters (mm).
Functional performance of Supine isometric chest lift test | Changes from baseline to 8 weeks when participants finish the intervention.
  The Supine Isometric Chest Lift Test will be used to assess the endurance of the abdominal muscles. Participants lie in a supine position and are instructed to lift the head and shoulders off the floor, maintaining the isometric position as long as possible. The holding time is recorded in seconds
Functional performance of Double Straight-Leg Raise Test | Changes from baseline to 8 weeks when participants finish the intervention.
  The Double Straight-Leg Raise Test will be used to assess the endurance of the trunk flexor muscles. Participants lie supine and are instructed to raise both legs to approximately 45 degrees and maintain this position as long as possible. The holding time is recorded in seconds
Functional performance of sorensen test | Changes from baseline to 8 weeks when participants finish the intervention.
  The Sorensen test will be used to assess the endurance of the back extensor muscles. Participants lie prone with the upper body extended beyond the edge of a table and are instructed to maintain a horizontal trunk position as long as possible. The total holding time is recorded in seconds
Functional performance of Active straight-leg raise fatigue task | Changes from baseline to 8 weeks when participants finish the intervention.
  Participants lifted the heel of the test leg to 20 cm for as long as possible. Participants were required to maintain pressure in the cuff beneath their back as close to 40 mm Hg as possible. Visual feedback of cuff pressure was provided throughout the task, but no instruction was given on how to affect cuff pressure. Task failure was defi ned as an inability to maintain heel height 10 cm or more off the plinth and/or a change in cuff pressure of 20 mm Hg or more.
Endurance of the pelvic stabilizing muscles | Changes from baseline to 8 weeks when participants finish the intervention.
  The manometry will provide measurements of pelvic floor muscle (PFM) function, including peak contraction pressure, average contraction pressure, and endurance capacity.
Functional performance of timed up and go test | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  Test instructions were given in Norwegian. Translated into English, the instructions were as follows: 'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
Functional performance of 6-Meter Walk Test | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  Subjects commenced the test in standing with their toes up against the tape marker. Test instructions translated into English were as follows: 'After "ready, set, go", walk as fast as you can up to the last white line without stopping or speaking along the way'. Performances were timed (to the nearest 100th of a second) between the 2m and 8m markers and later converted into speed in metres per second.
Functional performance of Four-Square Step Test | Changes from baseline to 8 weeks when participants finish the intervention.
  The Four-Square Step Test (FSST) will be used to assess dynamic balance and mobility. Participants are required to step rapidly in a specific sequence across four squares. The total time to complete the sequence is recorded in seconds.
Functional performance of Single-Leg Stance Test | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The Single-Leg Stance Test (SLST) will be used to assess static balance. Participants stand unassisted on one leg for as long as possible, with the test terminated when balance is lost or the non-supporting foot touches the ground. The holding time is recorded in seconds
Body composition | Changes from baseline to 8 weeks when participants finish the intervention.
  The InBody 770 bioelectrical impedance analysis (BIA) system will provide measurements of skeletal muscle mass (kg), lean body mass (kg), and total body water (L)
Body composition and bone mineral density | Changes from baseline to 8 weeks when participants finish the intervention.
  The dual-energy X-ray absorptiometry (DXA) system will provide measurements of bone mineral density (BMD) at the lumbar spine and hip regions (g/cm²)
Effectiveness of the app:System Usability Scale (SUS) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The System Usability Scale (SUS) will be used to evaluate the usability and user satisfaction of the system. The total score is converted to a 0-100 scale, where 0 represents the lowest usability and 100 represents the highest usability. Higher scores indicate better usability
Effectiveness of the app:Patient Satisfaction and Usability with Apps Questionnaire | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The Patient Satisfaction and Usability with Apps Questionnaire (pSUAPP) will be used to evaluate participants' satisfaction and perceived usability of the mobile health application. The total score ranges from 28 to 140 . Higher total scores indicate better user experience and app functionality
Self-perceived Change:Global Rating of Change Scale (GROC) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The Global Rating of Change Scale (GROC) rates perceived "overall change" on a 15-point Likert scale, with 7 (labeled "worse") on the left, +7 (labeled "better") on the right, and 0 in the middle (labeled "no change") compared to the baseline.
Quality of life and menopause related questionnaire:Brief Pain Inventory (BPI) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The Brief Pain Inventory (BPI) will be used to assess overall pain intensity and pain-related interference with daily activities. Each item is scored on a 0-10 scale.Higher scores represent worse outcomes.
Menopause related questionnaire:Menopause-Specific Quality of Life Questionnaire (MENQOL) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The Menopause-Specific Quality of Life Questionnaire (MENQOL) will provide domain-specific and overall scores assessing the impact of menopause on quality of life. The total score ranges from 0 to 174, with higher scores indicating worse symptoms and a greater negative impact on quality of life.
Quality of life and menopause related questionnaire:International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) will provide a total score (0-21) to evaluate the severity of urinary incontinence and its impact on quality of life, with higher scores indicating greater symptom severity.
Quality of life and menopause related questionnaire:Incontinence Quality of Life (I-QoL) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The Incontinence Quality of Life (I-QoL) questionnaire will assess quality of life related to urinary incontinence. Scores are transformed to a 0-100 scale. Higher scores indicate better incontinence-related quality of life
Quality of life and menopause related questionnaire:International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Changes from baseline to 8 weeks when participants finish the intervention, and follow-up assessments at 3 and 6 months post-intervention.
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be used to assess physical activity levels over the past 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No